CLINICAL TRIAL: NCT02656186
Title: Supplementation With Nutrients Modulating IGF-1 Negatively Correlated With Changes in the Levels of Proinflammatory Cytokines in Community-dwelling Elderly People at Risk of Undernutrition
Brief Title: Supplementation With Nutrients Modulating IGF-1 and Cytokines in Elderly People at Risk of Undernutrition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: YO_elderly
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm pretest-posttest (Experimental): In this study, the subjects served as their own controls. Subjects who were eligible based on inclusion criteria first entered into a 2-week pre-intervention period, during which they received nutrition counseling to keep their routine dietary habits. This was followed by an intervention period, during which an oral nutritional supplement was used over a period of 2 weeks.
  Interventions: Dietary Supplement: Pre-intervention; Dietary Supplement: Liquid nutritional supplement

INTERVENTIONS:
Dietary Supplement: Pre-intervention — First 2-weeks : keeping routine dietary habit
Dietary Supplement: Liquid nutritional supplement — Pre-intervention period was followed by an intervention period, during which consumed twice-daily 200 mL cartons of oral liquid nutritional supplementation (total 400 mL daily, containing 16 g protein, 12 g fat and 60 g carbohydrate and providing 400 kcal)

SUMMARY:
The purpose of this study was to determine the improvement in nutritional status, especially in the level of insulin-like growth factor-1 (IGF-1) and its relationship with changes in the circulating cytokine levels, after providing extra protein and energy contents to community-dwelling older adults at risk of undernutrition.

DETAILED DESCRIPTION:
Sixty of aged over 65 years, living independently in the community for elderly people, nondiabetic subjects with serum prealbumin of under 30 mg/dL and BMI under 25 kg/m2 were recruited. The subjects were followed for a 2-week pre-intervention period, followed by an intervention period, which they received 2 cartons of liquid oral nutritional supplementation daily for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily agree to participate and sign in informed consent form
* aged 65 years or older
* a serum prealbumin level≤30 mg/dL and a BMI<25 kg/m2

Exclusion Criteria:

* inability to perform oral ingestion
* known allergies to milk or eggs
* an inability to communicate, such as those with Alzheimer's disease
* malabsorption syndrome, a history of gastrectomy or enterectomy
* diabetes, liver disease, renal disease, neurological disease, pancreatitis, malignancy, cardiovascular or cerebrovascular disease, metabolic syndrome
* any other disease requiring treatment, medication or alcohol abuse
* any condition that the investigator believes may put the subjects at under risk

Ages: 65 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Prealbumin (mg/dL) | at pre-treatment (week -2)
Prealbumin (mg/dL) | at baseline (week 0)
Prealbumin (mg/dL) | at post-treatment (week 2)
Transferrin (mg/dL) | at pre-treatment (week -2)
Transferrin (mg/dL) | at baseline (week 0)
Transferrin (mg/dL) | at post-treatment (week 2)

SECONDARY OUTCOMES:
Weight (kg) | 4 weeks
  3 times during 4 weeks : at pre-treatment (week -2) / at baseline (week 0) / at post-treatment (week 2)
Body mass index (kg/m2) | 4 weeks
  3 times during 4 weeks : at pre-treatment (week -2) / at baseline (week 0) / at post-treatment (week 2)
Serum albumin (g/dL) | 4 weeks
  3 times during 4 weeks : at pre-treatment (week -2) / at baseline (week 0) / at post-treatment (week 2)
Insulin growth factor-1 (ng/mL) | 4 weeks
  3 times during 4 weeks : at pre-treatment (week -2) / at baseline (week 0) / at post-treatment (week 2)
Osmolality (mOsm/kgH2O) | 4 weeks
  3 times during 4 weeks : at pre-treatment (week -2) / at baseline (week 0) / at post-treatment (week 2)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D., Study Director — Department of Food & Nutrition, College of Human Ecology, Yonsei University 50 Yonsei-ro, Seodaemun-gu, Seoul, 03722, Korea

REFERENCES:
- [Derived] Kim M, Kim M, Lee YJ, Song HJ, Shim JK, Chang DH, Yu WK, Lee SH, Lee JH. Supplementation with nutrients modulating insulin-like growth factor-1 negatively correlated with changes in the levels of pro-inflammatory cytokines in community-dwelling elderly people at risk of undernutrition. J Hum Nutr Diet. 2017 Feb;30(1):27-35. doi: 10.1111/jhn.12447. Epub 2016 Dec 9. PMID 27933679